CLINICAL TRIAL: NCT03473314
Title: Open Label Prolonged-Use of Inhaled Gaseous Nitric Oxide (gNO) for a Single Adult With Non-Tuberculous Mycobacteria Infection
Brief Title: Prolonged-Use of Inhaled Gaseous Nitric Oxide (gNO) for Adult With Non-Tuberculous Mycobacteria Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Jeremy Road, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTM-SPU-01; H18-00512
Record Dates: First submitted 2018-03-14; First posted 2018-03-22 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Non-Tuberculous Mycobacterial Pneumonia
Keywords: Inhaled nitric oxide; Non-tuberculous mycobacteria; Drug resistant bacteria; Antimicrobial drug resistance

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nitric Oxide gas at 160ppm (Experimental): Nitric Oxide 160ppm for 50-80 minutes two -three times a day for 365 days
  Interventions: Drug: Nitric Oxide gas at 160ppm

INTERVENTIONS:
Drug: Nitric Oxide gas at 160ppm — Nitric oxide gas at 160 ppm inhaled three times daily for 50-80 min delivered with air as the carrier via inhalation for a maximum total of 90 days (extended 365 days twice). Total dose of 480 ppm hours per day.
  Other Names: Thiolanox

SUMMARY:
An open labeled Study (NCT03331445) is demonstrating encouraging safety and efficacy results for most subjects receiving 160ppm nitric oxide gas (gNO) for treatment of non-tuberculous mycobacteria (NTM) over a 15 day treatment regimen. In one subject, who had a reduction in sputum culture concentration of Bacterium bolletii from plus 3 to plus 1 corresponding to a 2-3 log10 cfu/gm reduction during the treatment, the one-week post treatment follow-up sputum culture had increased to plus 2. It is hypothesized that a longer treatment period may be necessary to fully eradicate NTM from the sputum culture in chronic lung disease. This study will extend the period of gNO exposure for a prolonged period of time (3 months) to attempt to fully eradicate the NTM in this single subject. This study will transition from the medical clinic to supervised delivery in the patient's home environment.

DETAILED DESCRIPTION:
Primary Objective: Determine the efficacy of prolonged delivery of inhaled nitric oxide to treat an adult patient with pulmonary NTM Primary Endpoint: Eradication of NTM growth in sputum cultures. Efficacy will be assessed by the antimicrobial effect of inhaled NO on the density of NTM species and other microorganisms in the sputum.

• as confirmed by measurement of semi-quantitative culture sputum growth which has been verified with serial dilution technique on Day 7, 14, 21 and every 21 days thereafter for 90 days as compared to pre-treatment baseline sputum culture.

Secondary Objective(s): Determine the safety & efficacy of inhaled nitric oxide

Secondary Endpoint(s):

1. Safety

   • as evaluated by the number of unanticipated adverse events during home delivery in clinical labs (hematology, coagulation, and serum chemistries); in vitals; in inspired concentration of NO, O2 and NO2 delivered to subject and; in methemoglobin and oxygen saturation levels.
2. Efficacy

   * as determined by improvement in lung function as measured by spirometry, endurance as measured by six minute walk-test and quality of life as determined by self-reporting quality of life questionnaire (CFQ-R) on Day 7, 14, 21 and every 21 days thereafter for 90 days as compared to pre-treatment baseline data.
   * as assessed by recurrence of NTM in sputum as confirmed by measurement of semi-quantitative culture sputum growth on Day 30 and 60 post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Has been previously diagnosed with NTM. [NTM defined as positive culture(s) of at least one species of Mycobacterium avium Complex (MAC) or Mycobacterium abscessus Complex (MABSC)]
* Has been previously treated with gNO for 15 days without complete eradication of NTM but with a decrease of at least 1-2 points on cultures.
* Male or female ≥19 years of age.
* Female not pregnant at time of study.
* Oxygen saturation on room air ≥92% at screening. (able to breathe without supplemental oxygen for 60 minutes)
* Non-smoker for at least 6 months prior to screening and agrees not to smoke during the study.
* Willing and able to comply with the treatment schedule and procedures.

Exclusion Criteria:

* History of frequent epistaxis (>1 episode/month)
* History of reactive pulmonary vascular hypertension
* Methemoglobin >3% at screening
* Liver function insufficiency aspartate aminotransferase/alanine aminotransferase (AST/ALT) >3 of normal values)
* Hemoglobin <10 g/dl
* Thrombocytopenia (platelet count <100,000/mm3) at screening
* Prothrombin time international ratio (INR) > 1.3 at screening
* On supplemental oxygen during gNO treatment (SaO2 < 90% for 50 minutes while resting in a chair).
* For women of child bearing potential:

  1. positive pregnancy test at screening or
  2. lactating or
  3. unwilling to practice a medically acceptable form of contraception from screening to Day 36 (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent)
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Eradication of NTM in sputum | 365 days
  The primary efficacy variable for this study is eradication of recovered NTM organisms in sputum colony forming unit (CFU) g (log 10) from baseline. Eradication will be defined as two negative sputum cultures post nitric oxide gas treatment over 60 days.

SECONDARY OUTCOMES:
Mean absolute change in forced expiratory volume at one second (FEV1)% from baseline. | 365 days
  Clinical Measurement of Mean absolute change in FEV1% from baseline to Day 365 (within group test).
Mean change in distance walked in the six-minute walk test from baseline | 365 days
  Clinical Measurement of Mean change in distance walked in the six-minute walk test from baseline.
Mean change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) scores for each domain from baseline | 365 days
  Clinical Measurement of Mean change in CFQ-R scores for each domain from baseline. Each domain measure the magnitude of severity for each of the 8 items. Respondents score each item using a 5-point likert scale ranging from 0 (no symptom) to 4 (the highest magnitude of severity). For item 1 (difficult to breathe), item 2 (feel feverish), item 3 (tired), item 6 (mucus), and item 7 (chest tightness) the response options are: 0=No symptom, 1=a little, 2=somewhat, 3=a good deal, 4=a great deal. For item 4 (chills/sweats), item 5 (cough), and item 8 (wheezing) the response options are: 0=no symptom, 1=slightly, 2=moderately, 3=very, 4=extremely.
Recurrence of NTM in sputum culture post NTM eradication. | 30 and 60 days post NTM eradication
  Measurement of recovered NTM organisms in sputum colony forming unit (CFU) g (log 10) post eradication. Eradication will be defined as two negative sputum cultures post nitric oxide gas treatment over 60 days.
Nitric oxide delivery effect on clinical values in home delivery | 365 days
  Safety measured as evaluated by the number of unanticipated adverse events in clinical labs (hematology, coagulation, and serum chemistries).
Nitric oxide delivery effect on key physiologic vital signs in home delivery | 365 days
  Safety measured as evaluated by the number of unanticipated adverse events in vitals signs (blood pressure, respiratory rate) and oxygen saturation levels during NO delivery.
Nitric oxide effect on delivery parameter concentrations in home delivery | 365 days
  Safety measured as evaluated by the number of unanticipated adverse events with inspired concentration of nitric oxide (NO), oxygen (O2) and nitrogen dioxide (NO2) delivered to subject.
Nitric oxide delivery effect on systemic methemoglobin levels in home delivery | 365 days
  Safety measured as evaluated by the number of unanticipated adverse events in pulseoixmetric arterial methemoglobin percent levels during nitric oxide delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Road, MD, Principal Investigator — University of British Columbia
Locations (1):
- Gordon Leslie Diamond Health Care Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided